CLINICAL TRIAL: NCT05021016
Title: An Open Study of the Safety, Reactogenicity and Immunogenicity of the Vaccine Based on Peptide Antigens for the Prevention of COVID-19 (EpiVacCorona), With the Involvement of Volunteers Aged 60 Years and Above (Phase III-IV)
Brief Title: Study of the EpiVacCorona Vaccine With the Involvement of Volunteers Aged 60 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: COV/pept-02/20
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: Covid19; SARS-CoV-2; EpiVacCorona; vaccination
MeSH Terms: conditions — COVID-19 | interventions — EpiVacCorona vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1: "Vaccine" (Experimental): 150 volunteers who will be vaccinated with the EpiVacCorona vaccine with two doses spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19)

INTERVENTIONS:
Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19) — The EpiVacCorona vaccine is intended to prevent COVID-19. The vaccine relies on chemically synthesized peptide antigens of SARS-CoV-2 proteins conjugated to a carrier protein and adsorbed on an aluminum-containing adjuvant (aluminum hydroxide).
  The vaccine induces the specific immunity against the SARS-CoV-2 coronavirus following two intramuscular injections spaced 21 to 28 days apart.
  The EpiVacCorona vaccine contributes to the development of protective immunity against SARS-CoV-2 coronavirus following two intramuscular administrations given 21 to 28 days apart.

SUMMARY:
The aim of the clinical study is to study the safety, reactogenicity and immunogenicity indicators of the EpiVacCorona vaccine, with the involvement of volunteers aged 60 years and above.

The research tasks are to:

* to evaluate the safety of the EpiVacCorona vaccine when administered twice intramuscularly, with the participation of volunteers aged 60 years and older;
* to evaluate the reactogenicity of the EpiVacCorona vaccine when administered twice intramuscularly, with the participation of volunteers aged 60 years and older;
* to identify any adverse effects to the administration of the vaccine;
* to study the humoral and cellular immune responses response following two doses of the EpiVacCorona vaccine, with the participation of volunteers aged 60 and older.

DETAILED DESCRIPTION:
The study will screen a maximum of 180 volunteers, of which it is proposed to include and randomize 150 men and women aged 60 years and older who meet the inclusion criteria and who do not have the exclusion criteria whose data will be used for subsequent safety and immunogenicity analysis.

The 150 volunteers will be vaccinated with the EpiVacCorona vaccine with two doses spaced 21 days apart, intramuscularly, at a dose of 0.5 ml.

The vaccine will be administered in procedure room settings only by a highly qualified specialist (vaccinator).

ELIGIBILITY:
Inclusion Criteria:

1. Availability of a signed and dated informed consent of the volunteer to participate in a clinical trial, prior to any of the study procedures.
2. Volunteers (men and women) aged 60 and above with stable indicators of basic vital functions.
3. Ability to attend all scheduled visits and all planned procedures and examinations.
4. Postmenopausal women over 60 years old.

Exclusion Criteria:

1. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS) or another coronavirus infection (HCoV-229E, HCOV-OC43, HCoV-NL63, HCoV-HKU1).
2. History of exposure to confirmed or suspected cases of SARS-CoV-2 infection within 1 month prior to randomization.
3. Positive for IgM or IgG to SARS-CoV-2 as detected during screening.
4. Positive PCR test for SARS-CoV-2 as detected during screening.
5. Clinically and laboratory (according to PCR data) confirmed disease caused by SARS-CoV-2 coronavirus, at the moment or in the past.
6. Serious post-vaccination reaction (body temperature above 40 °C , hyperemia or edema greater than 8 cm in diameter) or complication (collapse or shock-like state that developed within 48 hours after vaccination; convulsions, with or without of a febrile state) to a previous vaccination in the past.
7. Aggravated allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, history of serum disease, history of hypersensitivity or allergic reactions to the administration of any vaccines, any known allergic reactions to vaccine components, etc.).
8. History of Guillain-Barré syndrome (acute polyradiculitis).
9. Previous vaccination with rabies vaccines within less than 2 months prior to randomization, or planned vaccination with rabies vaccines within 1 month after immunization with the vaccine under study.
10. Hypersensitivity to any component of the product, allergy to vaccine components.
11. Persons in custody in detention facilities and those serving sentences in correctional facilities.
12. Symptoms of any disease at the time of inclusion in the study or if it has passed less than 4 weeks since recovery.
13. History of any acute respiratory illness less than 3 months prior to randomization.
14. Acute infectious or non-infectious diseases, exacerbation of chronic diseases less than 4 weeks prior to randomization.
15. History of tuberculosis (pulmonary and extrapulmonary), cancer, autoimmune diseases, skin diseases (pemphigus, psoriasis, eczema, atopic dermatitis).
16. Long-term use (more than 14 days) of immunosuppressants, systemic glucocorticosteroids or immunomodulatory drugs within 6 months prior to randomization.
17. Vaccination with any vaccine within one month prior to vaccination.
18. Use of immunoglobulin drugs or blood products within 3 months prior to randomization.
19. Acute or chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood, surgery on the gastrointestinal tract (except appendectomy).
20. Participation in other clinical trials less than 3 months prior to randomization.
21. Persons with alcohol or drug abuse (medications or narcotics). Use of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, or 200 ml of wine or 50 ml of alcohol) or history of alcoholism, narcomania or drug (medication) abuse.
22. Mental illness or neurasthenia.
23. Non-compliance with the inclusion criteria.
24. Positive test for HIV, viral hepatitis B and C, or syphilis.
25. Serious concomitant diseases or pathological conditions not listed above, which, according to the investigator's opinion, could complicate the assessment of the study results, including any pathological deviations from the age norms and laboratory norms of blood and urine parameters, clinically significant in the investigator's opinion.
26. Chronic diseases of the cardiovascular, bronchopulmonary, endocrine systems, gastrointestinal tract, liver, kidneys, blood, disease of the endocrine system in the exacerbation phase or that in the decompensation phase in the past or as detected during laboratory and imaging examination.

And:

1. The researcher's decision to exclude the volunteer for the benefit of the volunteer.
2. False inclusion (violation of inclusion and nonex-inclusion criteria) or the appearance of exclusion criteria during the study.
3. The decision of the researcher or the Sponsor to exclude the volunteer from the study due to a clinically significant deviation from the protocol/violation of the protocol.
4. Any undesirable phenomenon requiring the appointment of drugs not authorized by the protocol of this study.
5. Volunteer's refusal to continue his/her participation in the study or his/her lack of discipline.
6. Volunteer's desire to complete the study early for any reason.
7. Volunteer's failure to show up for a scheduled visit without the researcher's warning or loss of communication with the volunteer.
8. Positive urine drug test and / or positive alcohol breath test during the visit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of antibodies in virus neutralization reaction | 21 days after the second vaccination dose
  Geometric mean titer (GMT) of antibodies on day 21 following the second vaccination dose (Visit 17) in virus neutralization reaction

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of specific antibodies in ELISA | 21 days after the second vaccination dose
  The proportion of volunteers with increased levels of the immune response in terms of geometric mean titers of specific antibodies in ELISA is more than 4 times greater 21 days following the second vaccination dose
Specific neutralizing antibody titers in ELISA | 21 days after the second vaccination dose
  The proportion of volunteers with increased levels of the immune response in terms of specific neutralizing antibody titers in ELISA is more than 4 times greater 21 days following the second vaccination
The proportion of vaccinated volunteers with laboratory-confirmed SARS-CoV-2 symptoms in combination with one or more of the selected symptomsoV-2 symptoms in combination with one or more of the following symptoms | within 6 months following the first vaccination
  The proportion of vaccinated volunteers with laboratory-confirmed SARS-CoV-2 symptoms in combination with one or more of the following symptoms: fever or chills; cough; labored breathing or shortness of breath; fatigue; muscle pain; headache; loss of taste or smell; sore throat; nasal congestion or runny nose; nausea or vomiting; diarrhea within 6 months following vaccination
The proportion of volunteers with a T-cell response | 21 days after the second vaccination dose
  The proportion of volunteers with a T-cell response (CD4 +, CD8 +, CD4 + / CD8 +, concentration of interferon gamma, IL-2, IL-4) 21 days following the second vaccination dose
Geometric mean titers (GMT) of antibodies in the volunteers following vaccination and those in the convalescent volunteers vaccinated with the vaccine that recovered from COVID-19 | within 6 months following the first vaccination
  Geometric mean titers (GMT) of antibodies in the volunteers following vaccination and those in the convalescent volunteers vaccinated with the vaccine that recovered from COVID-19 of varying severity

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I. Kuzubov, PhD, Principal Investigator — FGBUZ MSCH-163, FMBA of Russia
Locations (1):
- Federal State Budgetary Institution of Healthcare "Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency" (FGBUZ MSCH-163, FMBA of Russia), Kol'tsovo, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No